CLINICAL TRIAL: NCT03302013
Title: Multi-center Clinical Study of Vanguard XP Bicruciate Knee System
Brief Title: All Ligaments Left In Knee Arthroplasty Trial
Acronym: ALLIKAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Zimmer Biomet (Industry); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11916; ISRCTN12584521 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2017-05-02; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Primary Osteoarthritis of Knee Nos
Keywords: Arthroplasty; Knee; Bicruciate retaining; Vanguard XP; Vanguard CR; Surgery; Zimmer Biomet; Joint Replacement; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vanguard XP Knee Replacement Surgery (Experimental): Participants randomised in this group will receive the Vanguard XP Bi-cruciate Retaining Knee Replacement System. This total knee replacement device (Vanguard XP) and surgical procedure retain the anterior cruciate ligament in the knee.
  Interventions: Procedure: Vanguard XP Bi-cruciate Retaining Knee Replacement System
- Vanguard CR Knee Replacement Surgery (Active Comparator): Participants randomised to this group will receive the Vanguard CR Single Cruciate Retaining Knee Replacement Surgery. This total knee replacement device (Vanguard CR) and surgical procedure sacrifice the anterior cruciate ligament and replaces it with artificial support. This is currently the standard practice for knee replacement surgery in the NHS.
  Interventions: Procedure: Vanguard CR Single Cruciate Retaining Knee System

INTERVENTIONS:
Procedure: Vanguard XP Bi-cruciate Retaining Knee Replacement System — Newer design of knee replacement retaining the Anterior Cruciate Ligament as well as the Posterior Cruciate Ligament.
  Arms: Vanguard XP Knee Replacement Surgery
Procedure: Vanguard CR Single Cruciate Retaining Knee System — Current 'gold standard' for total knee replacement which retains Posterior Cruciate Ligament but sacrifices the Anterior Cruciate Ligament, instead providing artificial support.
  Arms: Vanguard CR Knee Replacement Surgery

SUMMARY:
Compare the clinical and patient reported outcomes of the Vanguard XP Knee System to the Vanguard CR Knee System in patients with antero-medial osteoarthritis of the knee with an intact anterior cruciate ligament.

DETAILED DESCRIPTION:
The purpose of the proposed ALLIKAT study (All Ligaments Left in Knee Arthroplasty Trial) is to evaluate the early outcome of a Total Knee Replacement device that retains both cruciate (Vanguard XP) by comparing it with a control group of patients implanted with an established single cruciate retaining device (Vanguard CR). The study also aims to examine short and long term descriptive cohort outcome data. A small preference cohort group of 60 patients receiving the Vanguard XP Knee System will be recruited alongside the RCT group. This data will be used to confirm the external validity of the RCT group and to contribute to the safety data for the British Orthopaedic Association's Beyond Compliance Programme.

Evaluation will include intra-operative and post-operative complications, longer term survivorship and patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Primary Osteoarthritis of the knee involving one or more compartments of the joint.
* Intact Anterior and Posterior Cruciate Ligaments.
* Intact collateral ligaments.
* Correctable coronal deformity.
* No more than 15 degrees of fixed flexion deformity.

Exclusion Criteria:

* Age under 18 years.
* Revision knee replacement surgery.
* Rheumatoid Arthritis.
* Traumatic aetiology.
* History or clinical signs of ACL rupture.
* Previous arthroscopy related to ACL injury or reconstruction.
* Correction of a flexion contracture that may require extensive resection of distal femur.
* Altered pain perception and / or neurologic affection (for example as a complication arising from diabetes).
* Unable to consent for themselves.
* Patients with language or cognitive issues that may prevent them completing the follow up requirements.
* Contraindications for the device:

  * Cementless application of components.
  * BMI ≥40 kg/m2.
  * Use of Anterior Stabilized Bearings.
  * Patients with severe pre-operative varus or valgus deformity ≥ 15 degrees.
  * Correction or revision of previous joint replacement procedure on index knee.
  * Infection.
  * Sepsis.Osteomyelitis.
  * Osteoporosis (requiring treatment).
* Relative contraindications include:

  * Unco-operative patient or patient with neurologic disorders who is incapable of following directions.
  * Osteoporosis.
  * Metabolic disorders which may impair bone formation.
  * Osteomalacia.
  * Distant foci of infections which may spread to the implant site.
  * Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.
  * Vascular insufficiency, muscular atrophy, neuromuscular disease.
  * Incomplete or deficient soft tissue surrounding the knee, including the anterior cruciate ligament.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-09-05 (Actual); Primary Completion 2021-09-04 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score-Activity & Participation Questionnaire (OKS-APQ) | 3 years post randomisation
  Patient Reported Outcome Score - disease specific

SECONDARY OUTCOMES:
EQ-5D-3L | Post-operation (within 6 weeks); 1 & 3 years post randomisation
  Quality of Life Patient Reported Outcome Score
Forgotten Joint Score | Post operation (within 6 weeks), 1, 2 & 3 years post randomisation
  Patient Reported Outcome Score - disease specific
American Knee Society Score | Post operation (within 6 weeks), 1, 2 & 3 years post randomisation
  Functional Assessment of the knee
Complications | Post operation (within 6 weeks), 1 & 3 years post randomisation
  Adverse events and complications related to the knee surgery

OTHER OUTCOMES:
Radiographic Assessment | 1 & 3 Years Post Randomisation
  Evaluation of x-rays to assess Alignment, Radiolucency, Loosening, Fixation/Migration

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Price, Principal Investigator — University of Oxford
Locations (4):
- United Kingdom (4):
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham
  - North Bristol NHS Trust, Bristol
  - Frimley Health NHS Foundation Trust, Frimley

IPD SHARING:
Plan to Share IPD: No